CLINICAL TRIAL: NCT01564784
Title: AN OPEN-LABEL, RANDOMIZED PHASE 3 STUDY OF INOTUZUMAB OZOGAMICIN COMPARED TO A DEFINED INVESTIGATOR'S CHOICE IN ADULT PATIENTS WITH RELAPSED OR REFRACTORY CD22-POSITIVE ACUTE LYMPHOBLASTIC LEUKEMIA (ALL)
Brief Title: A Study Of Inotuzumab Ozogamicin Versus Investigator's Choice Of Chemotherapy In Patients With Relapsed Or Refractory Acute Lymphoblastic Leukemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B1931022; 2011-005491-41 (EudraCT Number)
Record Dates: First submitted 2012-03-26; First posted 2012-03-28 (Estimated); Results first posted 2018-01-17 (Actual); Last update posted 2019-01-09 (Actual); Status verified 2018-12

CONDITIONS: Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Inotuzumab Ozogamicin; fludarabine; Cytarabine; Granulocyte Colony-Stimulating Factor; Mitoxantrone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (Experimental)
  Interventions: Drug: inotuzumab ozogamicin
- Arm B (Active Comparator)
  Interventions: Drug: FLAG (fludarabine, cytarabine and G-CSF); Drug: HIDAC (high dose cytarabine); Drug: cytarabine and mitoxantrone

INTERVENTIONS:
Drug: inotuzumab ozogamicin — Dose: inotuzumab ozogamicin 0.8-0.5 mg/m^2 IV, weekly, 3 times per cycle Cycle length: 21-28 days Total number of cycles: 6
  Arms: Arm A
Drug: FLAG (fludarabine, cytarabine and G-CSF) — Dose: cytarabine 2.0 g/m^2/day IV days 1-6 fludarabine30 mg/m^2/day IV days 2-6 Cycle length: 28 days Total number of cycles: 4
  Arms: Arm B
Drug: HIDAC (high dose cytarabine) — cytarabine 3 g/m^2 IV every 12 hours for up to 12 times
  Arms: Arm B
Drug: cytarabine and mitoxantrone — mitoxantrone 12 mg/m^2 IV days 1-3 cytarabine 200 mg/m^2/day IV over 7 days cycle length: 15-20 days Total number of cycles: 4
  Arms: Arm B

SUMMARY:
This study will compare the efficacy, in terms of complete responses and overall survival, of inotuzumab ozogamicin versus investigator's choice of chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* CD22 expression
* Adequate liver and renal functions

Exclusion Criteria:

* Isolated extramedullary disease
* Active Central Nervous System [CNS] disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 326 (Actual)
Dates: Start 2012-08-02 (Actual); Primary Completion 2016-03-08 (Actual); Study Completion 2017-01-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (195):
- United States (94):
  - Investigational Drug Services - UC San Diego Moores Cancer Center, La Jolla, California
  - UC San Diego Medical Center - La Jolla, La Jolla, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Children's Center for Cancer and Blood Diseases, Childrens Hospital Los Angeles, Los Angeles, California
  - Keck Hospital of USC, Los Angeles, California
  - LAC+USC Medical Center, Los Angeles, California
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - USC/Norris Comprehensive Cancer Center / Investigational Drug Services, Los Angeles, California
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - UCLA Drug Information/Investigation Drug, Los Angeles, California
  - UCLA Hematology/Oncology Clinic, Los Angeles, California
  - UCLA Ronald Reagan Medical Center, Los Angeles, California
  - UCLA Rrmc, Los Angeles, California
  - UC Irvine Medical Center, Orange, California
  - Children's Hospital of Orange County, Orange, California
  - Freidenrich Center for Translational Research (CTRU), Stanford University, Palo Alto, California
  - UC San Diego Medical Center - Hillcrest, San Diego, California
  - Martha Hamilton, Investigational Drug Services, Dept of Pharmacy, Stanford, California
  - Stanford Cancer Institute, Stanford, California
  - Stanford University Hospital and Clinics, Stanford, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - University of Colorado Hospital, Cancer Center Infusion Center, Aurora, Colorado
  - University of Colorado Hospital, Aurora, Colorado
  - Yale-New Haven Hospital & Smilow Cancer Center, New Haven, Connecticut
  - Miami Children's Hospital, Miami, Florida
  - MD Anderson Cancer Center Orlando - 5th Floor Investigational Pharmacy, Orlando, Florida
  - MD Anderson Cancer Center Orlando, Orlando, Florida
  - Orlando Heart Health Institute, Orlando, Florida
  - Orlando Regional Medical Center, Orlando, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Investigational Drug Service, Emory University Clinic, Atlanta, Georgia
  - The Emory Clinic, Atlanta, Georgia
  - Winship Cancer Institute, Emory University, Atlanta, Georgia
  - Blood and Marrow Transplant Group of Georgia, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Georgia Regents Medical Center Pharmacy, Georgia Regents University Cancer Center, Augusta, Georgia
  - Georgia Regents University, Augusta, Georgia
  - Northwestern Medical Faculty Foundation, Chicago, Illinois
  - Northwestern Medicine Developmental Therapeutics Institute, Chicago, Illinois
  - Northwestern Memorial Hospital, Chicago, Illinois
  - The University of Chicago, Chicago, Illinois
  - University of Chicago Medical Center, Dept. of Pharmacy, Chicago, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kansas Hospital, Kansas City, Kansas
  - University of Kansas Cancer Center, Westwood, Kansas
  - Norton Cancer Institute, Louisville, Kentucky
  - Norton Cancer Institute, Suburban, Louisville, Kentucky
  - University of Maryland, Baltimore, Maryland
  - Oncology Investigational Drug Service, Baltimore, Maryland
  - The Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Massachusetts General Hospital (MGH), Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Health System-, Ann Arbor, Michigan
  - Karmanos Cancer Institute, Detroit, Michigan
  - Karmanos Cancer Institute Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Hackensack University Medical Center, Hackensack, New Jersey
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - University of New Mexico Comprehensive Cancer Center, Albuquerque, New Mexico
  - UNM Cancer Center, Albuquerque, New Mexico
  - Monter Cancer Center, Lake Success, New York
  - North Shore University Hospital, Manhasset, New York
  - New York Presbyterian Hospital-Weill Cornell Medical College, New York, New York
  - NewYork-Presbyterian Hospital, New York, New York
  - Weill Cornell Medical College - New York-Presbyterian Hospital, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Stony Brook University Medical Center, The Cancer Center, Stony Brook, New York
  - Division of Hematology/Oncology, Stony Brook University Hospital, Stony Brook, New York
  - UNC Cancer Hospital Infusion Pharmacy, Chapel Hill, North Carolina
  - UNC Hospitals - The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - OU Medical Center Presbyterian Tower, Oklahoma City, Oklahoma
  - Stephenson Cancer Center, Oklahoma City, Oklahoma
  - IDS-investigational drug pharmacy Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Penn State Milton S. Hershey Medical Center,, Hershey, Pennsylvania
  - Hollings Cancer Center, Charleston, South Carolina
  - MUSC Hospital, Charleston, South Carolina
  - Parkland Health and Hospital System, Dallas, Texas
  - Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - Baylor University Medical Center, Dallas, Texas
  - University of Texas Southwestern Universtiy Hospital - William P Clements Jr., Dallas, Texas
  - UT Southwestern Medical Center at Dallas, Dallas, Texas
  - UT Southwestern University Hospital- Zale Lipshy, Dallas, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - LDS Hospital, Salt Lake City, Utah
  - Seattle Cancer Care Alliance, Seattle, Washington
  - University of Washington, Seattle, Washington
  - West Virginia University Hospitals Pharmaceutical Services, Morgantown, West Virginia
  - West Virginia University Hospitals, Morgantown, West Virginia
- Sanatorio Allende, Córdoba, Argentina
- Australia (2):
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Eastern Clinical Research Unit, Box Hill Hospital, Box Hill, Victoria
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada
- China (7):
  - Guangdong General Hospital, Guangzhou, Guangdong
  - Henan Cancer Hostipal, Zhengzhou, Henan
  - The first hospital of jilin university, Changchun, Jilin
  - Beijing Chao-yang Hospital, Beijing
  - Peking University People's Hospital, Beijing
  - The 307th Hospital of PLA, Beijing
  - Institute of Hematology and Blood Diseases Hospital, Chinese Academy of Medical Sciences,, Tianjin
- Czechia (3):
  - Interni Hematologicka a Onkologicka Klinika, Brno
  - Fakultni Nemocnice Hradec Kralove, Hradec Králové
  - Fakultni nemocnice Kralovske Vinohrady, Prague
- Finland (2):
  - HUS-Kuvantaminen, Helsinki
  - HYKS/Hematologian klinikka, Helsinki
- France (10):
  - CHU de Dijon-Hopital d'Enfants-Service d'hematologie Clinique, Dijon
  - C.H.U. de Grenoble, Hopital Albert Michallon, Grenoble
  - Hopital Universitaire Andre Mignot, Le Chesnay
  - CHU Dupuytren, Limoges
  - Institut Paoli-Calmettes, Marseille
  - Hôpital Saint-Louis, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Institut de Cancérologie Lucien Neuwirth, Saint-Priest-en-Jarez
  - Iuct - Oncopole, Toulouse
  - CHU Brabois- Service d'hematologie, Vandœuvre-lès-Nancy
- Germany (7):
  - Zentralapotheke des Universitaetsklinikums Muenster, Münster, North Rhine-Westphalia
  - Universitätsklinikum Köln, Klinik I für Innere Medizin, Cologne
  - Klinikum der Goethe Universitaet, Frankfurt
  - Universitaetsklinikum Heidelberg, Heidelberg
  - Klinikum Rechts der Isar der TU München, München
  - Institut fuer klinische Radiologie, Münster
  - Universitaetsklinikum Muenster, Münster
- Hungary (2):
  - Egyesitett Szent Istvan és Szent Laszlo Korhaz-Rendelointezet;, Budapest
  - Debreceni Egyetem Orvos-es Egeszsegtudomanyi Centrum II. Belgyogyaszati Klinika, Debrecen
- Italy (26):
  - Azienda Ospedaliera Brotzu CTMO P.O. Businco, Cagliari, CA
  - Farmacia, Cagliari, CA
  - U.O. Radiodiagnostica, Cagliari, CA
  - IRST-Ematologia, Meldola (FC), FC
  - Istituto di Ematologia Seragnoli, Bologna
  - A.O.U. Vittorio Emanuele di Catania-Ospedale Ferrarotto, Catania
  - Radiology (Radiology Only), Catania
  - U.O. di Ematologia Dip. Medicine Specialistiche A.O.U. Arcispedale Sant'Anna, Cona, Ferrara
  - Clinica Ematologica, Genova
  - Pharmacy, Genova
  - Radiology Department (Radiology ONLY), Genova
  - Radiology Department, Genova
  - U.O. Ematologia 1, Genova
  - S.C. Pharmacy, Milan
  - S.C. Radiology, Milan
  - SC Ematologia, Milan
  - A.O. San Gerardo - Farmacia, Monza
  - A.O. San Gerardo di Monza, Monza
  - AORN "A. Cardarelli", Napoli
  - RAdiology Department (RAdiology only), Napoli
  - Clinica Ematologica, Pavia
  - Radiologist Department, Ravenna
  - Servizio di Farmacia, Ravenna
  - U.O. Ematologia, Ospedale S. Maria delle Croci, Ravenna
  - Clinica Ematologica, Udine
  - Radiology (Radiology Only), Udine
- Japan (8):
  - Nagoya Daini Red Cross Hospital, Nagoya, Aichi-ken
  - The Hospital of Hyogo College of Medicine, Nishinomiya-shi, Hyōgo
  - Tohoku University Hospital, Sendai, Miyagi
  - Osaka City University Hospital, Osaka, Osaka
  - National Cancer Center Hospital, Chuo-ku, Tokyo
  - Akita University Hospital, Akita
  - National Hospital Organization Kyushu Cancer Center, Fukuoka
  - Tokai University Hospital, Kanagawa
- Erasmus Medical Center, Rotterdam, South Holland, Netherlands
- Poland (4):
  - Klinika Hematologii i Transplantologii, Gdansk
  - Oddzial Hematologii, Klinika Hematologii, Regionalny Osrodek Onkologiczny Wojewodzki Szpital, Lodz
  - Instytut Hematologii i Transfuzjologii, Klinika Hematologii, Warsaw
  - Dolnoslaskie Centrum Transplantacji Komorkowych z Krajowym Bankiem Dawcow Szpiku, Wroclaw
- Singapore (2):
  - National University Hospital/National University Cancer Institute Singapore (NCIS), Singapore
  - Singapore General Hospital, Singapore
- South Korea (3):
  - Chonnam National University, Hwasun Hospital, Hwasun-Gun, Jeollanam-do
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (11):
  - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Universitario de Salamanca, Salamanca, Castille and LION
  - Hospital Vall d'Hebron, Barcelona, Catalonia
  - Hospital Son Llatzer, Palma de Mallorca, Mallorca
  - Hospital de la Santa Creu i Sant Pau(Nuevo Hospital), Barcelona
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Ramon y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital General Universitario Jose Maria Morales Meseguer, Murcia
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Clinico Universitario de Valencia, Valencia
- Sweden (2):
  - Universitetssjukhus Lund, Hematologkliniken, Lund
  - Hematology Center, Stockholm
- Taiwan (2):
  - Chang Gung Medical Foundation, Kaohsiung Branch, Kaohsiung City
  - National Taiwan University Hospital, Taipei
- United Kingdom (7):
  - Southampton General Hospital, Southampton, Hampshire
  - Bristol Haematology and Oncology Centre, Bristol
  - Castle Hill Hospital, Hull
  - Department of Academic Oncology, London
  - The Christie NHS Foundation Trust, Manchester
  - Nottingham University Hospitals NHS Trust, Nottingham
  - Churchill Hospital, Oxford

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Zhao Y, Laird AD, Roberts KG, Yafawi R, Kantarjian H, DeAngelo DJ, Stelljes M, Liedtke M, Stock W, Gokbuget N, O'Brien S, Jabbour E, Cassaday RD, Loyd MR, Olsen S, Neale G, Liu X, Vandendries E, Advani A, Mullighan CG. Association of leukemic molecular profile with efficacy of inotuzumab ozogamicin in adults with relapsed/refractory ALL. Blood Adv. 2024 Jun 25;8(12):3226-3236. doi: 10.1182/bloodadvances.2023012430. PMID 38607410
- [Derived] Stelljes M, Advani AS, DeAngelo DJ, Wang T, Neuhof A, Vandendries E, Kantarjian H, Jabbour E. Time to First Subsequent Salvage Therapy in Patients With Relapsed/Refractory Acute Lymphoblastic Leukemia Treated With Inotuzumab Ozogamicin in the Phase III INO-VATE Trial. Clin Lymphoma Myeloma Leuk. 2022 Sep;22(9):e836-e843. doi: 10.1016/j.clml.2022.04.022. Epub 2022 Apr 27. PMID 35643855
- [Derived] Shi Z, Zhu Y, Zhang J, Chen B. Monoclonal antibodies: new chance in the management of B-cell acute lymphoblastic leukemia. Hematology. 2022 Dec;27(1):642-652. doi: 10.1080/16078454.2022.2074704. PMID 35622074
- [Derived] Kantarjian HM, Stock W, Cassaday RD, DeAngelo DJ, Jabbour E, O'Brien SM, Stelljes M, Wang T, Paccagnella ML, Nguyen K, Sleight B, Vandendries E, Neuhof A, Laird AD, Advani AS. Inotuzumab Ozogamicin for Relapsed/Refractory Acute Lymphoblastic Leukemia in the INO-VATE Trial: CD22 Pharmacodynamics, Efficacy, and Safety by Baseline CD22. Clin Cancer Res. 2021 May 15;27(10):2742-2754. doi: 10.1158/1078-0432.CCR-20-2399. Epub 2021 Feb 18. PMID 33602684
- [Derived] Stock W, Martinelli G, Stelljes M, DeAngelo DJ, Gokbuget N, Advani AS, O'Brien S, Liedtke M, Merchant AA, Cassaday RD, Wang T, Zhang H, Vandendries E, Jabbour E, Marks DI, Kantarjian HM. Efficacy of inotuzumab ozogamicin in patients with Philadelphia chromosome-positive relapsed/refractory acute lymphoblastic leukemia. Cancer. 2021 Mar 15;127(6):905-913. doi: 10.1002/cncr.33321. Epub 2020 Nov 24. PMID 33231879
- [Derived] DeAngelo DJ, Advani AS, Marks DI, Stelljes M, Liedtke M, Stock W, Gokbuget N, Jabbour E, Merchant A, Wang T, Vandendries E, Neuhof A, Kantarjian H, O'Brien S. Inotuzumab ozogamicin for relapsed/refractory acute lymphoblastic leukemia: outcomes by disease burden. Blood Cancer J. 2020 Aug 7;10(8):81. doi: 10.1038/s41408-020-00345-8. PMID 32769965
- [Derived] Jabbour E, Gokbuget N, Advani A, Stelljes M, Stock W, Liedtke M, Martinelli G, O'Brien S, Wang T, Laird AD, Vandendries E, Neuhof A, Nguyen K, Dakappagari N, DeAngelo DJ, Kantarjian H. Impact of minimal residual disease status in patients with relapsed/refractory acute lymphoblastic leukemia treated with inotuzumab ozogamicin in the phase III INO-VATE trial. Leuk Res. 2020 Jan;88:106283. doi: 10.1016/j.leukres.2019.106283. Epub 2019 Nov 25. PMID 31790983
- [Derived] Fujishima N, Uchida T, Onishi Y, Jung CW, Goh YT, Ando K, Wang MC, Ono C, Matsumizu M, Paccagnella ML, Sleight B, Vandendries E, Fujii Y, Hino M. Inotuzumab ozogamicin versus standard of care in Asian patients with relapsed/refractory acute lymphoblastic leukemia. Int J Hematol. 2019 Dec;110(6):709-722. doi: 10.1007/s12185-019-02749-0. Epub 2019 Nov 13. PMID 31655984
- [Derived] Kantarjian HM, DeAngelo DJ, Stelljes M, Liedtke M, Stock W, Gokbuget N, O'Brien SM, Jabbour E, Wang T, Liang White J, Sleight B, Vandendries E, Advani AS. Inotuzumab ozogamicin versus standard of care in relapsed or refractory acute lymphoblastic leukemia: Final report and long-term survival follow-up from the randomized, phase 3 INO-VATE study. Cancer. 2019 Jul 15;125(14):2474-2487. doi: 10.1002/cncr.32116. Epub 2019 Mar 28. PMID 30920645
- [Derived] Jabbour EJ, DeAngelo DJ, Stelljes M, Stock W, Liedtke M, Gokbuget N, O'Brien S, Wang T, Paccagnella ML, Sleight B, Vandendries E, Advani AS, Kantarjian HM. Efficacy and safety analysis by age cohort of inotuzumab ozogamicin in patients with relapsed or refractory acute lymphoblastic leukemia enrolled in INO-VATE. Cancer. 2018 Apr 15;124(8):1722-1732. doi: 10.1002/cncr.31249. Epub 2018 Jan 30. PMID 29381191
- [Derived] Kebriaei P, Cutler C, de Lima M, Giralt S, Lee SJ, Marks D, Merchant A, Stock W, van Besien K, Stelljes M. Management of important adverse events associated with inotuzumab ozogamicin: expert panel review. Bone Marrow Transplant. 2018 Apr;53(4):449-456. doi: 10.1038/s41409-017-0019-y. Epub 2018 Jan 12. PMID 29330398
- [Derived] Kantarjian HM, DeAngelo DJ, Advani AS, Stelljes M, Kebriaei P, Cassaday RD, Merchant AA, Fujishima N, Uchida T, Calbacho M, Ejduk AA, O'Brien SM, Jabbour EJ, Zhang H, Sleight BJ, Vandendries ER, Marks DI. Hepatic adverse event profile of inotuzumab ozogamicin in adult patients with relapsed or refractory acute lymphoblastic leukaemia: results from the open-label, randomised, phase 3 INO-VATE study. Lancet Haematol. 2017 Aug;4(8):e387-e398. doi: 10.1016/S2352-3026(17)30103-5. Epub 2017 Jul 4. PMID 28687420
- [Derived] Kantarjian HM, DeAngelo DJ, Stelljes M, Martinelli G, Liedtke M, Stock W, Gokbuget N, O'Brien S, Wang K, Wang T, Paccagnella ML, Sleight B, Vandendries E, Advani AS. Inotuzumab Ozogamicin versus Standard Therapy for Acute Lymphoblastic Leukemia. N Engl J Med. 2016 Aug 25;375(8):740-53. doi: 10.1056/NEJMoa1509277. Epub 2016 Jun 12. PMID 27292104

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 164 participants were randomized to Inotuzumab Ozogamicin and 162 to Defined Investigator's Choice of Chemotherapy. Although only 143 participants were treated in the Defined Investigator's Choice of Chemotherapy arm, all 162 randomized participants were included in the intention-to-treat (ITT) population.
Groups:
- Inotuzumab Ozogamicin: Participants were treated with inotuzumab ozogamicin at a starting dose of 1.8 mg/m^2 (according to body surface area) per cycle with a divided-dose regimen using 3 weekly administrations. Participants received 0.8 mg/m^2/cycle on Week 1 (Day 1), followed by 0.5 mg/m^2 on Week 2 (Day 8) and Week 3 (Day 15) of a 21-day cycle, and administered as an intravenous infusion over 60 minutes. For participants who achieved a CR or CRi, or to allow recovery from toxicity, the length of Cycle 1 could be extended up to 28 days (ie, 1 week treatment-free interval starting on Day 21). For participants who achieved CR or CRi, the inotuzumab ozogamicin dose administered on Week 1 was reduced to 0.5 mg/m^2 (for a total cycle dose of 1.5 mg/m^2/cycle) for Cycles 2 through 6 (maximum number of cycles permitted). For Cycles 2 through 6, the cycle length was 28 days for all participants (regardless of remission status).
- Defined Investigator's Choice of Chemotherapy: Participants received fludarabine, cytarabine, granulocyte-colony stimulating factor (FLAG), mitoxantrone + cytarabine (MXN/Ara-C), or high-dose cytarabine (HIDAC), according to the Investigator's choice.
Period: Overall Study
Arm/Group | Inotuzumab Ozogamicin | Defined Investigator's Choice of Chemotherapy
Started | 164 (Treated (164 randomized)) | 143 (Treated (162 randomized))
Completed | 30 | 10
Not Completed | 134 | 133
Not completed — Other | 1 | 0
Not completed — Subject refused further follow-up | 1 | 6
Not completed — Lost to Follow-up | 1 | 1
Not completed — Death | 131 | 126

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Inotuzumab Ozogamicin | Defined Investigator's Choice of Chemotherapy | Total
Number analyzed (Participants) | 164 | 143 | 307
Age, Continuous [Mean (Standard Deviation); unit: Years] | 45.9 (17.07) | 45.6 (16.32) | 45.7 (16.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73 | 51 | 124
  Male | 91 | 92 | 183

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Hematologic Remission (Complete Remission [CR]/Complete Remission With Incomplete Hematologic Recovery [CRi]) as Assessed by the Endpoint Adjudication Committee (EAC)
Description: CR was the disappearance of leukemia indicated by less than (<) 5 percent (%) marrow blasts & absence of peripheral blood leukemic blasts, with recovery of hematopoiesis defined by absolute neutrophil count (ANC) greater than or equal to (≥)1000 per microliter (/μL) & platelets ≥100,000/μL. C1 extramedullary disease status (i.e. complete disappearance of measurable & non-measurable extramedullary disease with the following exceptions: for participants with at least 1 measurable lesion, all nodal masses greater than (>) 1.5 centimeters (cm) in greatest transverse diameter (GTD) at baseline must have regressed to less than or equal to (≤) 1.5 cm in GTD; all nodal masses ≥1 cm & ≤1.5 cm in GTD at baseline must have regressed to <1 cm GTD or reduced by 75% in sum of products of greatest diameters, no new lesions, spleen & other previously enlarged organs must have regressed in size & must not be palpable) was required. CRi was defined as CR except ANC <1000/μL &/or platelets <100,000/μL.
Time Frame: Screening, Day 16 to 28 of Cycles 1, 2 and 3, then every 1 to 2 cycles (or as clinically indicated) up to approximately 4 weeks (end of treatment [EoT]) from the last dose
Population: ITT218 population - included the ITT population (all participants randomized) for the initial 218 participants.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Inotuzumab Ozogamicin | Defined Investigator's Choice of Chemotherapy
Number analyzed (Participants) | 109 | 109
Percentage of Participants | 80.7 [72.1 to 87.7] | 29.4 [21.0 to 38.8]
Statistical Analysis 1: Comparison: Inotuzumab Ozogamicin vs Defined Investigator's Choice of Chemotherapy; Test type: Superiority or Other; p < 0.0001, 1-sided p-value based on Chi-square test; If any cell count was <5, p-value was based on Fisher's exact test; Rate difference = 51.4, 97.5% CI 2-sided [38.4 to 64.3]

2. Primary Outcome: Overall Survival (OS)
Description: OS was defined as the time from randomization to date of death due to any cause. Participants last known to be alive were censored at date of last contact.
Time Frame: Up to 5 years after randomization or 2 years from randomization of the last participant, whichever occurs first.
Population: ITT population - included all participants randomized. Although only 143 participants were treated in the Defined Investigator's Choice of Chemotherapy arm, all 162 randomized participants were included in the ITT population.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Inotuzumab Ozogamicin | Defined Investigator's Choice of Chemotherapy
Number analyzed (Participants) | 164 | 162
Months | 7.7 [6.0 to 9.2] | 6.2 [4.7 to 8.3]
Statistical Analysis 1: Comparison: Inotuzumab Ozogamicin vs Defined Investigator's Choice of Chemotherapy; Test type: Superiority or Other; p = 0.0105, 1-sided stratified log-rank p-value; Hazard Ratio (HR) = 0.751, 97.5% CI 2-sided [0.568 to 0.993] — Stratified HR, i.e., based on analysis stratified by randomization stratification factors

3. Secondary Outcome: Duration of Remission (DoR) for Participants Who Achieved CR/CRi (Per Investigator Assessment)
Description: DoR was defined as time from date of first response in responders (CR/CRi per Investigator assessment) to date of PFS event (i.e. death, progressive disease [objective progression, relapse from CR/CRi or treatment discontinuation due to global deterioration of health status] or starting new induction therapy or post-therapy stem cell transplant [SCT] without achieving CR/CRi). Responders without PFS events were censored at the last valid disease assessment including follow-up.
Time Frame: Up to 2 years from randomization
Population: Participants in the ITT218 population who achieved CR/CRi
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Inotuzumab Ozogamicin | Defined Investigator's Choice of Chemotherapy
Number analyzed (Participants) | 85 | 32
Months | 5.4 [4.3 to 8.0] | 3.5 [2.2 to 6.6]
Statistical Analysis 1: Comparison: Inotuzumab Ozogamicin vs Defined Investigator's Choice of Chemotherapy; Test type: Superiority or Other; p = 0.0021, 1-sided stratified log-rank p-value; Hazard Ratio (HR) = 0.490, 95% CI 2-sided [0.297 to 0.809] — Stratified HR, i.e., based on analysis stratified by randomization stratification factors

4. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS was defined as time from date of randomization to earliest date of the following events: death, progressive disease (objective progression, relapse from CR/CRi or treatment discontinuation due to global deterioration of health status) and starting new induction therapy or post-therapy SCT without achieving CR/CRi. Participants without a PFS event at time of analysis were censored at the last valid disease assessment. In addition, participants with documentation of an event after an unacceptably long interval (>28 weeks if there was post-baseline disease assessment, or >12 weeks if there was no post-baseline assessment) since the previous disease assessment were censored at the time of the previous assessment (date of randomization if no post-baseline assessment). Post-study treatment follow-up disease assessments was included. Kaplan-Meier method used and 2-sided 95% confidence interval (CI) calculated based on the Brookmeyer and Crowley method.
Time Frame: Up to 2 years from randomization
Population: ITT population. Although only 143 participants were treated in the Defined Investigator's Choice of Chemotherapy arm, all 162 randomized participants were included in the ITT population.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Inotuzumab Ozogamicin | Defined Investigator's Choice of Chemotherapy
Number analyzed (Participants) | 164 | 162
Months | 5.0 [3.9 to 5.8] | 1.7 [1.4 to 2.1]
Statistical Analysis 1: Comparison: Inotuzumab Ozogamicin vs Defined Investigator's Choice of Chemotherapy; Test type: Superiority or Other; p < 0.0001, 1-sided stratified log-rank p-value; Hazard Ratio (HR) = 0.450, 97.5% CI 2-sided [0.336 to 0.602] — Stratified HR, i.e., based on analysis stratified by randomization stratification factors

5. Secondary Outcome: Percentage of Participants Who Had a Hematopoietic Stem-Cell Transplant (HSCT)
Description: HSCT rate was defined as the percentage of participants who underwent SCT following treatment with inotuzumab ozogamicin or Investigator's choice of chemotherapy.
Time Frame: Up to 19 weeks from last dose
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Inotuzumab Ozogamicin | Defined Investigator's Choice of Chemotherapy
Number analyzed (Participants) | 164 | 162
Percentage of Participants | 42.7 [35.0 to 50.6] | 11.1 [6.7 to 17.0]
Statistical Analysis 1: Comparison: Inotuzumab Ozogamicin vs Defined Investigator's Choice of Chemotherapy; Test type: Superiority or Other; p < 0.0001, 1-sided p-value based on Chi-square test; If any cell count was <5, p-value was based on Fisher's exact test; Rate difference = 31.6, 95% CI 2-sided [22.6 to 40.6]

6. Secondary Outcome: Percentage of Participants Achieving MRD Negativity (Based on Central Laboratory Analysis) in Participants Achieving a CR/CRi (Per EAC Assessment)
Description: MRD analysis was performed at least once in participants with prior assessment of CR or CRi. Bone marrow aspirates, collected at screening and during the study, were sent to the central laboratory and analyzed using multiparametric flow cytometry. The antibody combinations were designed to maximize discrimination between normal and abnormal cells of B-cell lineage and similar maturational stage and included antibodies detecting cluster of differentiation (CD) 9, CD10, CD13, CD19, CD20, CD33, CD34, CD38, CD45, CD58, CD66c, and CD123. A peripheral blood sample was provided if a participant had an inadequate bone marrow aspirate at screening. MRD negativity was considered to have been achieved if the lowest value of MRD from the first date of CR/CRi to EoT was <1 × 10^-4 blasts/nucleated cells.
Time Frame: Up to approximately 4 weeks (EoT) from last dose of study drug
Population: Participants in the ITT218 population achieving CR/CRi (per EAC Assessment)
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Inotuzumab Ozogamicin | Defined Investigator's Choice of Chemotherapy
Number analyzed (Participants) | 88 | 32
Percentage of Participants | 78.4 [68.4 to 86.5] | 28.1 [13.7 to 46.7]
Statistical Analysis 1: Comparison: Inotuzumab Ozogamicin vs Defined Investigator's Choice of Chemotherapy; Test type: Superiority or Other; p < 0.0001, 1-sided p-value based on Chi-Square test; If any cell count is <5, p-value was based on Fisher's exact test

7. Secondary Outcome: Cytogenetic Status (Based on Local Laboratory Analysis) of Participants With CR/CRi (Per EAC Assessment)
Description: Karyotyping was required locally, at screening and at least once during the study in participants who had abnormal cytogenetics at baseline and who achieved CR/CRi. Data presented below are for participants who achieved CR/CRi per EAC and had abnormal karyotype at screening.
Time Frame: Up to approximately 4 weeks (EoT) from last dose of study drug
Population: Participants in the ITT218 population who had abnormal cytogenetics at baseline and who achieved CR/CRi
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Inotuzumab Ozogamicin | Defined Investigator's Choice of Chemotherapy
Number analyzed (Participants) | 54 | 22
Percentage of Participants | 3.7 [0.5 to 12.7] | 18.2 [5.2 to 40.3]
Statistical Analysis 1: Comparison: Inotuzumab Ozogamicin vs Defined Investigator's Choice of Chemotherapy; Abnormal at Screening; Test type: Superiority or Other; p = 0.3168, 1-sided p-value based on Chi-Square test; If any cell count is <5, p-value was based on Fisher's exact test
Statistical Analysis 2: Comparison: Inotuzumab Ozogamicin vs Defined Investigator's Choice of Chemotherapy; Abnormal after remission; Test type: Superiority or Other; p = 0.2160, 1-sided p-value based on Chi-Square test; If any cell count is <5, p-value was based on Fisher's exact test

8. Secondary Outcome: Maximum Observed Inotuzumab Ozogamicin Serum Concentration (Cmax) and Pre-Dose Inotuzumab Ozogamicin Serum Concentration (Ctrough) Following Single and Multiple Dosing
Description: Blood samples were collected and analyzed for inotuzumab ozogamicin serum concentrations using a validated high performance liquid chromatography with tandem mass spectrometry (HPLC/MS/MS) method with a lower limit of quantification of 1.0 nanograms per milliliter (ng/mL). Cmax was the maximum observed concentration occurring between 0-8 hours post-dose. Ctrough was the concentration prior to subsequent dose (pre-dose) occurring after 8 hours. n = number of observations (non-missing concentrations).
Time Frame: Days 1, 4, 8, and 15 of Cycle 1, Days 1 and 8 of Cycle 2 and Day 1 of Cycle 4
Population: Pharmacokinetic (PK) evaluable population - included all participants with available PK data.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Inotuzumab Ozogamicin
Number analyzed (Participants) | 163
ng/mL
  Cmax (Cycle 1 Day 1, 1 hour post-dose) (n=128) | 211 (232)
  Ctrough (Cycle 4 Day 1, pre-dose) (n=46) | 57.9 (29.8)
  Cmax (Cycle 4 Day 1, 1 hour post-dose) (n=37) | 308 (362)

9. Secondary Outcome: Change From Baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire, Core 30 (EORTC QLQ-C30) Score
Description: This questionnaire comprised 30 questions within which are 9 multi-item scales & 6 single-item measures. There are 5 functional scales; physical, role, cognitive, emotional & social, 3 symptom scales; fatigue, pain, & nausea & vomiting, & a global health status/quality of life (QoL) scale. There are 5 single item measures assessing additional symptoms commonly reported by cancer patients (loss of appetite, insomnia, constipation, diarrhea, & dyspnea) & a single item concerning perceived financial impact of the disease. Most questions used a 4 point scale (1='not at all' to 4='very much'); 2 questions used a 7-point scale (1='very poor' to 7='excellent'). Scores were averaged & transformed to a scale ranging from 0 to 100; a higher score indicates a better level of functioning or greater degree of symptoms.
Time Frame: Day 1 of each cycle prior to dosing and EoT
Population: as for outcome 4
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Inotuzumab Ozogamicin | Defined Investigator's Choice of Chemotherapy
Number analyzed (Participants) | 164 | 162
Score on a scale
  Physical Functioning C2D1 | 0.48 (1.53) | 0.32 (3.55)
  Physical Functioning C3D1 | 3.15 (1.97) | -13.33 (7.70)
  Physical Functioning C4D1 | 5.33 (2.84) | 0.00 (NA) — n=1
  Physical Functioning C5D1 | 11.52 (3.51) | NA (NA) — n=0
  Physical Functioning C6D1 | 7.22 (5.94) | NA (NA) — n=0
  Physical Functioning EoT | -3.38 (2.03) | -8.17 (2.67)
  Role Functioning C2D1 | 5.45 (2.79) | -1.59 (8.21)
  Role Functioning C3D1 | 11.81 (3.19) | -11.11 (5.56)
  Role Functioning C4D1 | 16.67 (5.47) | 0.00 (NA) — n=1
  Role Functioning C5D1 | 12.88 (6.10) | NA (NA) — n=0
  Role Functioning C6D1 | 16.67 (11.42) | NA (NA) — n=0
  Role Functioning EoT | 1.32 (3.59) | -12.37 (4.09)
  Emotional Functioning C2D1 | 5.21 (1.76) | 4.76 (6.77)
  Emotional Functioning C3D1 | 7.41 (1.85) | -19.44 (10.02)
  Emotional Functioning C4D1 | 5.69 (1.63) | 0.00 (NA) — n=1
  Emotional Functioning C5D1 | 6.82 (2.83) | NA (NA) — n=0
  Emotional Functioning C6D1 | 2.78 (4.27) | NA (NA) — n=0
  Emotional Functioning EoT | -0.91 (1.80) | 4.35 (2.96)
  Cognitive Functioning C2D1 | 4.05 (1.47) | 0.00 (3.98)
  Cognitive Functioning C3D1 | 5.79 (2.11) | -5.56 (14.70)
  Cognitive Functioning C4D1 | 4.58 (2.86) | 16.67 (NA) — n=1
  Cognitive Functioning C5D1 | 0.76 (4.17) | NA (NA) — n=0
  Cognitive Functioning C6D1 | -8.33 (2.51) | NA (NA) — n=0
  Cognitive Functioning EoT | 0.83 (1.82) | 0.54 (2.89)
  Social Functioning C2D1 | 4.20 (2.46) | -2.38 (7.21)
  Social Functioning C3D1 | 5.56 (3.25) | -27.78 (20.03)
  Social Functioning C4D1 | 10.42 (4.95) | 0.00 (NA) — n=1
  Social Functioning C5D1 | 12.88 (6.00) | NA (NA) — n=0
  Social Functioning C6D1 | 16.67 (5.03) | NA (NA) — n=0
  Social Functioning EoT | 1.82 (2.84) | -2.15 (4.78)
  Global Health Status C2D1 | 3.98 (2.03) | 0.40 (4.62)
  Global Health Status C3D1 | 9.38 (3.15) | -16.67 (12.73)
  Global Health Status C4D1 | 11.25 (3.69) | 8.33 (NA) — n=1
  Global Health Status C5D1 | 8.71 (6.68) | NA (NA) — n=0
  Global Health Status C6D1 | 0.69 (6.76) | NA (NA) — n=0
  Global Health Status EoT | 0.00 (2.83) | -0.40 (3.28)
  Dyspnoea C2D1 | -5.41 (2.72) | -7.94 (6.47)
  Dyspnoea C3D1 | -7.41 (3.24) | 11.11 (11.11)
  Dyspnoea C4D1 | -12.50 (4.25) | 0.00 (NA) — n=1
  Dyspnoea C5D1 | -3.03 (6.55) | NA (NA) — n=0
  Dyspnoea C6D1 | -2.78 (6.43) | NA (NA) — n=0
  Dyspnoea EoT | -2.31 (3.09) | 0.54 (3.95)
  Insomnia C2D1 | -2.40 (3.01) | 1.59 (5.85)
  Insomnia C3D1 | -9.26 (3.38) | 0.00 (19.25)
  Insomnia C4D1 | -7.50 (3.27) | 0.00 (NA) — n=1
  Insomnia C5D1 | -4.55 (4.55) | NA (NA) — n=0
  Insomnia C6D1 | -11.11 (9.48) | NA (NA) — n=0
  Insomnia EoT | -2.31 (3.09) | 0.00 (3.91)
  Appetite Loss C2D1 | -4.20 (2.83) | 3.17 (7.24)
  Appetite Loss C3D1 | -8.33 (4.31) | 0.00 (0.00)
  Appetite Loss C4D1 | -11.67 (5.54) | 0.00 (NA) — n=1
  Appetite Loss C5D1 | -6.06 (7.80) | NA (NA) — n=0
  Appetite Loss C6D1 | 2.78 (9.59) | NA (NA) — n=0
  Appetite Loss EoT | -1.32 (3.54) | 11.83 (4.41)
  Constipation C2D1 | -1.21 (2.47) | 0.00 (5.14)
  Constipation C3D1 | 0.47 (3.44) | 0.00 (0.00)
  Constipation C4D1 | -2.50 (3.66) | 0.00 (NA) — n=1
  Constipation C5D1 | 0.00 (5.37) | NA (NA) — n=0
  Constipation C6D1 | 5.56 (5.56) | NA (NA) — n=0
  Constipation EoT | 2.64 (2.60) | -0.54 (2.71)
  Diarrhoea C2D1 | -3.30 (2.17) | -1.59 (4.87)
  Diarrhoea C3D1 | -5.09 (2.61) | -11.11 (11.11)
  Diarrhoea C4D1 | -0.83 (3.27) | 0.00 (NA) — n=1
  Diarrhoea C5D1 | -9.52 (4.68) | NA (NA) — n=0
  Diarrhoea C6D1 | -2.78 (4.95) | NA (NA) — n=0
  Diarrhoea EoT | 2.31 (1.89) | 3.76 (3.35)
  Financial Difficulties C2D1 | -1.80 (1.99) | 0.00 (8.72)
  Financial Difficulties C3D1 | 0.47 (3.24) | 0.00 (0.00)
  Financial Difficulties C4D1 | -1.67 (3.37) | 0.00 (NA) — n=1
  Financial Difficulties C5D1 | -3.03 (3.74) | NA (NA) — n=0
  Financial Difficulties C6D1 | -5.56 (3.75) | NA (NA) — n=0
  Financial Difficulties EoT | 0.33 (3.09) | 2.19 (2.80)
  Fatigue C2D1 | -4.10 (2.40) | 5.82 (6.88)
  Fatigue C3D1 | -8.33 (3.02) | 22.22 (6.42)
  Fatigue C4D1 | -9.17 (4.64) | -11.11 (NA) — n=1
  Fatigue C5D1 | -7.32 (5.61) | NA (NA) — n=0
  Fatigue C6D1 | 0.00 (6.42) | NA (NA) — n=0
  Fatigue Eot | -0.33 (2.66) | 5.73 (3.27)
  Nausea and Vomiting C2D1 | 0.15 (2.16) | -0.79 (2.69)
  Nausea and Vomiting C3D1 | -4.63 (2.80) | 0.00 (0.00)
  Nausea and Vomiting C4D1 | -3.33 (3.17) | -16.67 (NA) — n=1
  Nausea and Vomiting C5D1 | 2.27 (2.96) | NA (NA) — n=0
  Nausea and Vomiting C6D1 | 0.00 (2.90) | NA (NA) — n=0
  Nausea and Vomiting EoT | -0.17 (2.33) | 3.49 (2.43)
  Pain C2D1 | -8.86 (2.71) | -7.14 (7.68)
  Pain C3D1 | -8.56 (3.73) | -5.56 (14.70)
  Pain C4D1 | -4.17 (3.81) | -33.33 (NA) — n=1
  Pain C5D1 | 0.76 (7.48) | NA (NA) — n=0
  Pain C6D1 | -2.78 (9.59) | NA (NA) — n=0
  Pain EoT | -1.98 (2.88) | -7.26 (3.75)
Statistical Analysis 1: Comparison: Inotuzumab Ozogamicin vs Defined Investigator's Choice of Chemotherapy; Physical Functioning; Test type: Superiority or Other; p = 0.0139, Mixed Models Analysis; Treatment, time, treatment-by-time interaction, and baseline included as covariate; Mean Difference (Net) = 6.9, 95% CI 2-sided [1.4 to 12.3]
Statistical Analysis 2: Comparison: Inotuzumab Ozogamicin vs Defined Investigator's Choice of Chemotherapy; Role Functioning; Test type: Superiority or Other; p = 0.0065, Mixed Models Analysis; Treatment, time, treatment-by-time interaction, and baseline included as covariate; Mean Difference (Net) = 11.4, 95% CI 2-sided [3.2 to 19.5]
Statistical Analysis 3: Comparison: Inotuzumab Ozogamicin vs Defined Investigator's Choice of Chemotherapy; Emotional Functioning; Test type: Superiority or Other; p = 0.3307, Mixed Models Analysis; Treatment, time, treatment-by-time interaction, and baseline included as covariate; Mean Difference (Net) = -2.3, 95% CI 2-sided [-6.9 to 2.3]
Statistical Analysis 4: Comparison: Inotuzumab Ozogamicin vs Defined Investigator's Choice of Chemotherapy; Cognitive Functioning; Test type: Superiority or Other; p = 0.1904, Mixed Models Analysis; Treatment, time, treatment-by-time interaction, and baseline included as covariate; Mean Difference (Net) = 2.8, 95% CI 2-sided [-1.4 to 7.0]
Statistical Analysis 5: Comparison: Inotuzumab Ozogamicin vs Defined Investigator's Choice of Chemotherapy; Social Functioning; Test type: Superiority or Other; p = 0.0336, Mixed Models Analysis; Treatment, time, treatment-by-time interaction, and baseline included as covariate; Mean Difference (Net) = 8.4, 95% CI 2-sided [0.7 to 16.1]
Statistical Analysis 6: Comparison: Inotuzumab Ozogamicin vs Defined Investigator's Choice of Chemotherapy; Global Health Status; Test type: Superiority or Other; p = 0.1572, Mixed Models Analysis; Treatment, time, treatment-by-time interaction, and baseline included as covariate; Mean Difference (Net) = 4.3, 95% CI 2-sided [-1.7 to 10.3]
Statistical Analysis 7: Comparison: Inotuzumab Ozogamicin vs Defined Investigator's Choice of Chemotherapy; Dyspnoea; Test type: Superiority or Other; p = 0.1281, Mixed Models Analysis; Treatment, time, treatment-by-time interaction, and baseline included as covariate; Mean Difference (Net) = -4.7, 95% CI 2-sided [-10.8 to 1.4]
Statistical Analysis 8: Comparison: Inotuzumab Ozogamicin vs Defined Investigator's Choice of Chemotherapy; Insomnia; Test type: Superiority or Other; p = 0.6207, Mixed Models Analysis; Treatment, time, treatment-by-time interaction, and baseline included as covariate; Mean Difference (Net) = -1.7, 95% CI 2-sided [-8.7 to 5.2]
Statistical Analysis 9: Comparison: Inotuzumab Ozogamicin vs Defined Investigator's Choice of Chemotherapy; Appetite Loss; Test type: Superiority or Other; p = 0.0193, Mixed Models Analysis; Treatment, time, treatment-by-time interaction, and baseline included as covariate; Mean Difference (Net) = -8.7, 95% CI 2-sided [-16.0 to -1.4]
Statistical Analysis 10: Comparison: Inotuzumab Ozogamicin vs Defined Investigator's Choice of Chemotherapy; Constipation; Test type: Superiority or Other; p = 0.6249, Mixed Models Analysis; Treatment, time, treatment-by-time interaction, and baseline included as covariate; Mean Difference (Net) = 1.4, 95% CI 2-sided [-4.4 to 7.3]
Statistical Analysis 11: Comparison: Inotuzumab Ozogamicin vs Defined Investigator's Choice of Chemotherapy; Diarrhoea; Test type: Superiority or Other; p = 0.1534, Mixed Models Analysis; Treatment, time, treatment-by-time interaction, and baseline included as covariate; Mean Difference (Net) = -3.0, 95% CI 2-sided [-7.2 to 1.1]
Statistical Analysis 12: Comparison: Inotuzumab Ozogamicin vs Defined Investigator's Choice of Chemotherapy; Financial Difficulties; Test type: Superiority or Other; p = 0.4915, Mixed Models Analysis; Treatment, time, treatment-by-time interaction, and baseline included as covariate; Mean Difference (Net) = -2.5, 95% CI 2-sided [-9.7 to 4.7]
Statistical Analysis 13: Comparison: Inotuzumab Ozogamicin vs Defined Investigator's Choice of Chemotherapy; Fatigue; Test type: Superiority or Other; p = 0.1789, Mixed Models Analysis; Treatment, time, treatment-by-time interaction, and baseline included as covariate; Mean Difference (Net) = -4.4, 95% CI 2-sided [-10.8 to 2.0]
Statistical Analysis 14: Comparison: Inotuzumab Ozogamicin vs Defined Investigator's Choice of Chemotherapy; Nausea and Vomiting; Test type: Superiority or Other; p = 0.4578, Mixed Models Analysis; Treatment, time, treatment-by-time interaction, and baseline included as covariate; Mean Difference (Net) = -1.6, 95% CI 2-sided [-6.0 to 2.7]
Statistical Analysis 15: Comparison: Inotuzumab Ozogamicin vs Defined Investigator's Choice of Chemotherapy; Pain; Test type: Superiority or Other; p = 0.8428, Mixed Models Analysis; Treatment, time, treatment-by-time interaction, and baseline included as covariate; Mean Difference (Net) = -0.7, 95% CI 2-sided [-7.3 to 6.0]

10. Secondary Outcome: Change From Baseline in EuroQol 5 Dimension Health Questionnaire (EQ-5D) Index Score
Description: The EQ-5D self-report questionnaire is a standardized measure of health status developed by the EuroQoL Group. It consists of the EQ-5D descriptive system and a visual analogue scale (VAS), EQ-VAS. The EQ-5D descriptive system measures a participants' health state on 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 3 levels, reflecting "no problems", "some problems", and "extreme problems". The EQ-VAS records the respondent's self-rated health on a scale from 0 (worst imaginable health state) to 100 (best imaginable health state); higher scores indicate a better health state. EQ-5D summary index is obtained with a formula that weights each level of the dimensions. The index-based score is interpreted along a continuum of 0 (death) to 1 (perfect health).
Time Frame: Day 1 of each cycle prior to dosing and EoT
Population: as for outcome 4
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Inotuzumab Ozogamicin | Defined Investigator's Choice of Chemotherapy
Number analyzed (Participants) | 164 | 162
Score on a scale
  Cycle 2, Day 1 | 0.00 (0.02) | 0.02 (0.03)
  Cycle 3, Day 1 | 0.01 (0.02) | -0.08 (0.08)
  Cycle 4, Day 1 | 0.04 (0.03) | 0.00 (NA) — n=1
  Cycle 5, Day 1 | 0.04 (0.04) | NA (NA) — n=0
  Cycle 6, Day 1 | 0.03 (0.04) | NA (NA) — n=0
  EoT | -0.01 (0.02) | -0.04 (0.02)
Statistical Analysis 1: Comparison: Inotuzumab Ozogamicin vs Defined Investigator's Choice of Chemotherapy; Test type: Superiority or Other; p = 0.1710, Mixed Models Analysis; Treatment, time, treatment-by-time interaction, and baseline included as covariate; Mean Difference (Net) = 0.03, 95% CI 2-sided [-0.01 to 0.07]

11. Secondary Outcome: Change From Baseline in EQ-5D VAS
Description: The EQ-5D self-report questionnaire is a standardized measure of health status developed by the EuroQoL Group. It consists of the EQ-5D descriptive system and a visual analogue scale (VAS), EQ-VAS. The EQ-5D descriptive system measures a participants' health state on 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 3 levels, reflecting "no problems", "some problems", and "extreme problems". The EQ-VAS records the respondent's self-rated health on a scale from 0 (worst imaginable health state) to 100 (best imaginable health state); higher scores indicate a better health state.
Time Frame: Day 1 of each cycle prior to dosing and EoT
Population: as for outcome 4
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Inotuzumab Ozogamicin | Defined Investigator's Choice of Chemotherapy
Number analyzed (Participants) | 164 | 162
Score on a scale
  Cycle 2, Day 1 | 5.81 (2.14) | 5.90 (4.21)
  Cycle 3, Day 1 | 8.13 (2.53) | 19.67 (17.80)
  Cycle 4, Day 1 | 7.13 (3.37) | 44.00 (NA) — n=1
  Cycle 5, Day 1 | 7.62 (4.43) | NA (NA) — n=0
  Cycle 6, Day 1 | 15.09 (9.14) | NA (NA) — n=0
  EoT | 4.62 (2.38) | -0.52 (2.88)
Statistical Analysis 1: Comparison: Inotuzumab Ozogamicin vs Defined Investigator's Choice of Chemotherapy; Test type: Superiority or Other; p = 0.1172, Mixed Models Analysis; Treatment, time, treatment-by-time interaction, and baseline included as covariate; Mean Difference (Net) = 4.6, 95% CI 2-sided [-1.2 to 10.4]

12. Secondary Outcome: Percentage of Participants With Veno-Occlusive Liver Disease (VOD)/Sinusoidal Obstruction Syndrome (SOS) Following Post Study HSCT
Description: VOD/SOS was defined as the occurrence of 2 out of the following 3 clinical criteria: 1) total serum bilirubin level >34 micromoles per liter (μmol/L) (>2.0 milligrams per deciliter [mg/dL]), 2) an increase in liver size from baseline or development of right upper quadrant pain of liver origin and 3) sudden weight gain >2.5% (eg, within a 72 hour period) because of fluid accumulation in the weeks following infusion of study drug or chemotherapy, or HSCT conditioning/preparative therapy, or development of ascites not present at baseline following such exposures AND the absence of other explanations for these signs and symptoms, OR development of bilirubin elevation, weight gain, or hepatomegaly plus histologic abnormalities on liver biopsy demonstrating hepatocyte necrosis in zone 3 of the liver acinus, sinusoidal fibrosis, and centrilobular hemorrhage, with or without fibrosis of the terminal hepatic venules.
Time Frame: Up to 2 years from randomization
Population: Participants in the Safety population with post-study HSCT. A site visit in July 2017 (after clinical database lock), confirmed a fourth case of VOD/SOS occurred in the Defined Investigators Choice of Chemotherapy arm in March 2013 (approximately 3 months after the last dose).This was not entered on the CRF and therefore, is not included below.
Measure: Number; unit: Percentage of Participants
Arm/Group | Inotuzumab Ozogamicin | Defined Investigator's Choice of Chemotherapy
Number analyzed (Participants) | 79 | 35
Percentage of Participants | 22.8 | 8.6

ADVERSE EVENTS:
Time Frame: SAEs and non-serious AEs are summarized from Cycle 1 Day 1 up to 42 days after last dose, or any time after Cycle 1 Day1 (treatment-related).
Description: An event may appear as both an AE & SAE. However, what is presented are distinct events. An event may be categorized as serious in 1 participant & non-serious in another participant, or 1 participant may have experienced both a serious & non-serious event. Events were reported up to at least 28 days after last dose.
Arm/Group | Inotuzumab Ozogamicin | Defined Investigator's Choice of Chemotherapy
Serious Adverse Events (participants affected / at risk) | 85/164 | 72/143
Other Adverse Events (participants affected / at risk) | 159/164 | 143/143
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Inotuzumab Ozogamicin (N=164) | Defined Investigator's Choice of Chemotherapy (N=143)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 19 | 27
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Left ventricular dysfunction (Cardiac disorders) | 2 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Pericarditis (Cardiac disorders) | 1 | 0
Blindness unilateral (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 1
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 0
Colitis ischaemic (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1
Gastritis haemorrhagic (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Ileal perforation (Gastrointestinal disorders) | 0 | 1
Intestinal ischaemia (Gastrointestinal disorders) | 1 | 1
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 1 | 0
Large intestinal ulcer (Gastrointestinal disorders) | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Mesenteric haemorrhage (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 0
Oesophageal stenosis (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 2 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 3 | 0
Chest pain (General disorders) | 1 | 0
Disease progression (General disorders) | 8 | 5
Fatigue (General disorders) | 1 | 0
Mucosal inflammation (General disorders) | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 2 | 2
Pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 5 | 3
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Hepatic vein thrombosis (Hepatobiliary disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 3
Venoocclusive liver disease (Hepatobiliary disorders) | 23 | 3 — After clinical database lock, a fourth case of VOD/SOS was confirmed in the Defined Investigators Choice of Chemotherapy arm in March 2013 (approximately 3 months after last dose). This was not entered on the CRF and therefore, is not included below.
Adenoviral upper respiratory infection (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1
Bacteraemia (Infections and infestations) | 3 | 1
Bacterial infection (Infections and infestations) | 0 | 1
Brain abscess (Infections and infestations) | 1 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 0 | 1
Candida infection (Infections and infestations) | 1 | 1
Cellulitis (Infections and infestations) | 1 | 1
Clostridium difficile colitis (Infections and infestations) | 2 | 1
Clostridium difficile infection (Infections and infestations) | 1 | 0
Corona virus infection (Infections and infestations) | 1 | 0
Cytomegalovirus chorioretinitis (Infections and infestations) | 0 | 1
Device related infection (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0
Enteritis necroticans (Infections and infestations) | 0 | 1
Enterococcal bacteraemia (Infections and infestations) | 1 | 0
Enterococcal sepsis (Infections and infestations) | 1 | 0
Escherichia bacteraemia (Infections and infestations) | 2 | 2
Escherichia sepsis (Infections and infestations) | 1 | 2
Febrile infection (Infections and infestations) | 1 | 0
Fungaemia (Infections and infestations) | 1 | 0
Fungal infection (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 2 | 0
Klebsiella bacteraemia (Infections and infestations) | 0 | 1
Klebsiella infection (Infections and infestations) | 0 | 1
Liver abscess (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 1 | 2
Necrotising fasciitis fungal (Infections and infestations) | 0 | 1
Neutropenic sepsis (Infections and infestations) | 3 | 4
Parainfluenzae virus infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 10 | 0
Pneumonia fungal (Infections and infestations) | 0 | 3
Pneumonia pseudomonal (Infections and infestations) | 0 | 1
Pseudomonal bacteraemia (Infections and infestations) | 1 | 2
Pseudomonal sepsis (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 4 | 10
Septic embolus (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 3 | 3
Serratia bacteraemia (Infections and infestations) | 1 | 0
Sinusitis fungal (Infections and infestations) | 1 | 0
Staphylococcal bacteraemia (Infections and infestations) | 1 | 1
Staphylococcal sepsis (Infections and infestations) | 2 | 1
Systemic candida (Infections and infestations) | 1 | 1
Systemic mycosis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 1
Urinary tract infection fungal (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 3
Fluid overload (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 1 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Bone infarction (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 1 | 1
Headache (Nervous system disorders) | 2 | 0
Nervous system disorder (Nervous system disorders) | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 2 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pharyngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 6
Respiratory tract oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 3
Shock haemorrhagic (Vascular disorders) | 1 | 0
Thrombophlebitis (Vascular disorders) | 0 | 1
Mucormycosis (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Inotuzumab Ozogamicin (N=164) | Defined Investigator's Choice of Chemotherapy (N=143)
Anaemia (Blood and lymphatic system disorders) | 54 | 79
Febrile neutropenia (Blood and lymphatic system disorders) | 27 | 52
Leukopenia (Blood and lymphatic system disorders) | 47 | 54
Lymphopenia (Blood and lymphatic system disorders) | 31 | 36
Neutropenia (Blood and lymphatic system disorders) | 79 | 66
Thrombocytopenia (Blood and lymphatic system disorders) | 80 | 86
Tachycardia (Cardiac disorders) | 6 | 16
Dry eye (Eye disorders) | 1 | 8
Abdominal distension (Gastrointestinal disorders) | 10 | 2
Abdominal pain (Gastrointestinal disorders) | 19 | 26
Abdominal pain upper (Gastrointestinal disorders) | 11 | 12
Constipation (Gastrointestinal disorders) | 28 | 34
Diarrhoea (Gastrointestinal disorders) | 30 | 55
Dyspepsia (Gastrointestinal disorders) | 3 | 9
Nausea (Gastrointestinal disorders) | 52 | 68
Stomatitis (Gastrointestinal disorders) | 5 | 9
Vomiting (Gastrointestinal disorders) | 25 | 35
Asthenia (General disorders) | 14 | 14
Chest pain (General disorders) | 3 | 9
Chills (General disorders) | 18 | 17
Fatigue (General disorders) | 41 | 24
Mucosal inflammation (General disorders) | 6 | 19
Oedema peripheral (General disorders) | 13 | 13
Pain (General disorders) | 12 | 8
Pyrexia (General disorders) | 49 | 57
Hyperbilirubinaemia (Hepatobiliary disorders) | 35 | 23
Bacteraemia (Infections and infestations) | 4 | 13
Pneumonia (Infections and infestations) | 4 | 12
Sinusitis (Infections and infestations) | 4 | 8
Contusion (Injury, poisoning and procedural complications) | 10 | 3
Fall (Injury, poisoning and procedural complications) | 11 | 4
Alanine aminotransferase increased (Investigations) | 25 | 18
Aspartate aminotransferase increased (Investigations) | 37 | 16
Blood alkaline phosphatase increased (Investigations) | 21 | 10
Gamma-glutamyltransferase increased (Investigations) | 35 | 12
Lipase increased (Investigations) | 15 | 1
White blood cell count decreased (Investigations) | 10 | 9
Decreased appetite (Metabolism and nutrition disorders) | 19 | 18
Fluid overload (Metabolism and nutrition disorders) | 2 | 8
Hyperglycaemia (Metabolism and nutrition disorders) | 11 | 12
Hypoalbuminaemia (Metabolism and nutrition disorders) | 10 | 7
Hypocalcaemia (Metabolism and nutrition disorders) | 11 | 15
Hypokalaemia (Metabolism and nutrition disorders) | 25 | 33
Hypomagnesaemia (Metabolism and nutrition disorders) | 10 | 12
Hyponatraemia (Metabolism and nutrition disorders) | 5 | 9
Hypophosphataemia (Metabolism and nutrition disorders) | 9 | 10
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 16 | 10
Bone pain (Musculoskeletal and connective tissue disorders) | 3 | 10
Pain in extremity (Musculoskeletal and connective tissue disorders) | 13 | 16
Dizziness (Nervous system disorders) | 12 | 16
Headache (Nervous system disorders) | 45 | 38
Anxiety (Psychiatric disorders) | 8 | 11
Depression (Psychiatric disorders) | 4 | 9
Insomnia (Psychiatric disorders) | 24 | 22
Cough (Respiratory, thoracic and mediastinal disorders) | 22 | 23
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 | 18
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 24 | 12
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 | 10
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 8
Erythema (Skin and subcutaneous tissue disorders) | 7 | 9
Pruritus (Skin and subcutaneous tissue disorders) | 8 | 10
Rash (Skin and subcutaneous tissue disorders) | 14 | 27
Hypertension (Vascular disorders) | 9 | 8
Hypotension (Vascular disorders) | 12 | 22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 60 days from the time submitted to the sponsor for review. Investigators will, on request, remove any previously undisclosed Confidential Information (other than the Study results themselves) before disclosure.